CLINICAL TRIAL: NCT04668898
Title: Dissecting Oligogenic Biomarkers in Ashkenazi Jews With Parkinson's Disease
Brief Title: LRRK2, GBA and Other Genetic Biomarkers in Eastern European (Ashkenazi) Jews With and Without Parkinson's Disease
Acronym: BioPD
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Rachel Saunders-Pullman, Professor, Neurology, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-1846; 1U01NS107016-01A1 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; LRRK2; GBA Gene Mutation
Keywords: Parkinson's disease; Parkinsonian Disorders; LRRK2; GBA; Movement Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The study team will be collecting DNA (ACD tubes), serum, plasma, RNA, peripheral blood monocytes, and urine. In a select group of patients, the study team will be collecting cerebrospinal fluid through a lumbar puncture. Samples are deposited in the Parkinson's Disease Biomarker Program repository.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- LRRK2 Parkinson Disease: Individuals with LRRK2-related Parkinson Disease
- GBA Parkinson Disease: Individuals with GBA-related Parkinson Disease
- Idiopathic Parkinson Disease: Individuals with Idiopathic (without any known genetic cause) Parkinson Disease
- LRRK2 non-manifesting carriers: Individuals without Parkinson Disease who have a LRRK2 mutation
- GBA non-manifesting carriers: Individuals without Parkinson Disease who have a GBA mutation
- Healthy control: Individuals without a personal or family history (1st or 2nd degree) of a neurodegenerative disease

SUMMARY:
Single site observational study focused on elucidating the genes and biochemical pathways involved in causing Parkinson disease.

DETAILED DESCRIPTION:
This single site study, is enrolling Parkinson disease (PD) patients and their family members and is limited to participants of Ashkenazi (Eastern European) Jewish descent with GBA and LRRK2 mutations, or with 3 or more family members with PD. Follow-up will be for three years. Participants must be in the New York City area yearly and willing to come to Mount Sinai Downtown for yearly 2 hour study visits which include obtaining personal medical and family history information, blood, urine and spinal fluid samples, neurological exam and neuropsychiatric testing. De-identified data and samples will be securely stored at a central NIH-run repository for access by other researchers. Spinal fluid collection is encouraged but optional.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease patients and their family members and is limited to participants of Ashkenazi (Eastern European) Jewish descent with GBA and LRRK2 mutations, or with 3 or more family members with PD
* Participants must be local to the New York City area and willing to come to Mount Sinai Downtown for annual 2 hour study visits which include obtaining personal medical and family history information, blood, urine and spinal fluid samples, neurological exam and neuropsychiatric testing. Spinal fluid collection is encouraged but optional.

Exclusion Criteria:

-Patients who do not have Parkinson disease or family members of Ashkenazi (Eastern European) Jewish descent who either has a GBA or LRRK2 mutations OR who has 3 or more family members with PD.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson disease patients and their family members who are of Ashkenazi (Eastern European) Jewish descent who either have a GBA or LRRK2 mutations or who have 3 or more family members with PD.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Elucidate blood-based genetic biomarkers in Parkinson's disease | five years
  Discovery and validation of new blood-based genetic biomarkers (both DNA and expression-based) for Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Saunders-Pullman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Laurie Ozelius, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mount Sinai-- Downtown Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Clinical data deposited in Parkinson Disease Biomarker Program DMR after study visit
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. The type of analysis will be for individual participant data meta-analysis. Data are available indefinitely at: https://pdbp-demo.cit.nih.gov/researchers.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04668898/ICF_000.pdf